CLINICAL TRIAL: NCT00476112
Title: A Phase II/III Prospective, Randomized, Double-Blind, Placebo-Controlled, Multi-Centred Tolerance and Efficacy Study of RSD1235 in Patients With Atrial Flutter
Brief Title: A Phase II/III Tolerance and Efficacy Study of RSD1235 in Patients With Atrial Flutter
Acronym: Scene 2
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Advanz Pharma (Industry)
Collaborators: Astellas Pharma US, Inc. (Industry)
Responsible Party: Sheila Grant, VP of Product Development, Vernakalant, Cardiome Pharma Corp.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1235-0703B
Record Dates: First submitted 2007-05-18; First posted 2007-05-21 (Estimated); Last update posted 2008-04-02 (Estimated); Status verified 2008-03

CONDITIONS: Atrial Flutter
Keywords: Atrial flutter; RSD1235
MeSH Terms: conditions — Atrial Flutter | interventions — vernakalant

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Atrial flutter duration of 3 hours to <45 days
  Interventions: Drug: Vernakalant Injection 20 mg/mL

INTERVENTIONS:
Drug: Vernakalant Injection 20 mg/mL
  Other Names: RSD1235; Vernakalant; Vernakalant Injection; Vernakalant (iv)

SUMMARY:
This study will attempt to demonstrate the effectiveness of RSD1235 in the conversion of atrial flutter (AFL) to sinus rhythm.

DETAILED DESCRIPTION:
There are approximately 2 million reported prevalent cases of atrial fibrillation and atrial flutter (AFL) in the United States (Heart Disease & Stroke Statistics - 2003 Update, AHA). These arrhythmias may be occasional or sustained. AF/AFL is usually associated with age, and general physical condition, rather than with a specific cardiac event, as is often the case with ventricular arrhythmia. While not directly fatal, these arrhythmias cause discomfort and can lead to stroke or congestive heart failure.

This Phase II/III trial is Cardiome's first study with RSD1235 for the treatment of atrial flutter. The study seeks to demonstrate RSD1235's abilities to convert AFL to sinus rhythm. The patient population will have atrial flutter of duration greater than 3 hours and less than or equal to 45 days.

This is a double-blind, placebo-controlled, randomized study in patients with AFL; stratification will be based on duration of AFL. Treatment will be considered successful if there is a treatment-induced conversion of atrial arrhythmia to sinus rhythm for a minimum of 1-minute by Hour 1.5 (Time 0 = start of first infusion). All patients will be evaluated for safety.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Have an atrial arrhythmia with dysrhythmic symptoms that has been sustained for greater than 3 hours and up to 45 days.
* Have adequate anticoagulant therapy.

Exclusion Criteria:

* Have a QRS > 0.14 s unless patient has pacemaker or uncorrected QT > 0.440 seconds as measured on a 12-lead ECG.
* Be concurrently participating in another drug study or have received an investigational drug within 30 days prior to enrollment, or have previously received RSD1235.
* Have serious diseases/illnesses that could interfere with the conduct or validity of the study or compromise patient safety.
* Have received IV Class I or Class III antiarrhythmic drugs or IV amiodarone within 24 hours prior to dosing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2003-08; Primary Completion 2004-09 (Actual); Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
To demonstrate the effectiveness of RSD1235 in the conversion of AFL to sinus rhythm. Treatment will be considered successful if there is treatment-induced conversion of AFL to sinus rhythm for a minimum of 1 minute duration by Hour 1.5. | The proportion of patients with atrial flutter who have treatment-induced conversion of atrial flutter to sinus rhythm for a minimum duration of one minute in the first 90 minutes after the first exposure to study treatment.

SECONDARY OUTCOMES:
To assess the safety of RSD1235 in this patient population and to assess the efficacy of RSD1235 in lowering the ventricular response rate in patients with AFL. | Treatment-induced reduction of the ventricular response rate within 50 minutes of first exposure to treatment for patient with atrial flutter.

CONTACTS AND LOCATIONS:
Overall Officials: Sheila Grant, MBA, Study Director — Advanz Pharma
Locations (24):
- United States (5):
  - Regional Cardiology Associates, Sacramento, California
  - Thoracic and Cardiovascular Institute, Lansing, Michigan
  - Medical College of Virginia, Richmond, Virginia
  - McGuire VA Medical Center, Richmond, Virginia
  - Marshfield Clinic, Marshfield, Wisconsin
- Canada (8):
  - Heart Health Institute, Rockyview General Hospital, Calgary, Alberta
  - University of Calgary, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Hamilton Health Sciences, Hamilton General Hospital, Hamilton, Ontario
  - Ottawa Hospitals (Civic & General), Ottawa, Ontario
  - Institut de Cardiologie de Montreal, Montreal, Quebec
  - Hopital Notre-Dame du CHUM, Montreal, Quebec
  - CHUM-Hotel-Dieu de Montreal, Montreal, Quebec
- Denmark (9):
  - Aalborg University, Aalborg
  - H:S Bispebjerg Hospital, Copenhagen
  - Centralsygehuset Esbjerg Varde, Esbjerg
  - Glostrup Amtssygehus, Glostrup Municipality
  - Gentofte Amtssygehus, Hellerup
  - Herlev Amtssygehus, Kardiologisk, Herlev
  - Sygehus Vendsyssel Hjorring, Hjørring
  - Holstebro centralsygehus, Holstebro
  - Hvidovre Hospital, Kardiologisk, Hvidovre
- Sweden (2):
  - Universitetssjukhuset MAS, Malmo
  - Centrallasarettet, Vasteras, Västerås

REFERENCES:
- [Derived] Camm AJ, Toft E, Torp-Pedersen C, Vijayaraman P, Juul-Moller S, Ip J, Beatch GN, Dickinson G, Wyse DG; Scene 2 Investigators. Efficacy and safety of vernakalant in patients with atrial flutter: a randomized, double-blind, placebo-controlled trial. Europace. 2012 Jun;14(6):804-9. doi: 10.1093/europace/eur416. Epub 2012 Jan 29. PMID 22291438